CLINICAL TRIAL: NCT03642106
Title: Reducing Alcohol, Tobacco, and Drug Use Among Latino Immigrant Youth: A Preliminary Test of the ¡Unidos Se Puede! Program
Brief Title: Unidos Against ATOD Use Intervention Trial
Acronym: TWC
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Oklahoma State University (Other)
Collaborators: National Institute of General Medical Sciences (NIGMS) (NIH); National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Principal Investigator, Ronald Cox, Professor, Oklahoma State University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: IRB-21-290; 5P20GM109097-02 (NIH); 1R15DA049232-01 (NIH)
Record Dates: First submitted 2018-04-13; First posted 2018-08-22 (Actual); Last update posted 2022-07-27 (Actual); Status verified 2022-07

CONDITIONS: Substance Use
Keywords: Adolescent; Latino; Immigrant
MeSH Terms: conditions — Substance-Related Disorders

STUDY DESIGN:
Intervention Model Description: To accomplish the mentioned aims, we propose an attention placebo randomized control trial. For this trial, we will recruit a sample of youth and their parents (N=120 dyads) from a random sample of Latino 6th and 7th grade students in Tulsa Public Schools. Those meeting the inclusion/exclusion criteria and agreeing to participate will provide baseline data before being randomly assigned to either the treatment or control condition (n=60 dyads each).
  Participants will be followed for 12 months post-baseline, during which time we will collect psychosocial measures annually near the end of each school year (May to June). The study will collect psychosocial measures from parents and youth.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Unidos Se Puede (Active Comparator): Unidos Se Puede: consists of 5-weekly Family Workshops, 6 monthly booster sessions, 10-months success coaching, adolescent group activities and will be compared to an attention placebo control.
  Interventions: Behavioral: Unidos Se Puede
- Attention placebo control (Placebo Comparator): Placebo consists of after school club for youth.
  Interventions: Behavioral: Unidos Se Puede

INTERVENTIONS:
Behavioral: Unidos Se Puede — The intervention consists of: (1) encouraging parental involvement in child schooling, general parenting skills, and coping strategies ; (2) fostering child social emotional learning (SEL) through assigning a near-peer success coach to help develop critical thinking, problem solving, and goal setting skills; and (3) promoting positive peer affiliations through participation in regular activities that facilitate bonding to prosocial institutions.
  Other Names: UWC

SUMMARY:
Adolescent alcohol tobacco and drug (ATOD) use is a major public health concern, with rates for Latino middle school youth higher than other ethnic groups. One well-established precursor of adolescent ATOD use is psychosocial stress. The proposed project examines the preliminary efficacy of Unidos to decrease ATOD use among Latino youth in new settlement areas. The goals of this efficacy trial will be achieved by accomplishing two specific aims: (1) Evaluate the potential of the intervention to delay the initiation into or reduce ATOD use among Latino youth who are 1st to 2nd generation immigrants; and (2) Evaluate the intervention's ability to strengthen known protective factors against ATOD use among adolescents-specifically child personal agency and parent-child, peer, and school relationships.

The study's primary hypothesis is: The Unidos Se Puede program will delay initiation of ATOD use of current non-users and reduce use among current users.

DETAILED DESCRIPTION:
Adolescent alcohol tobacco and drug (ATOD) use is a major public health concern, with rates for Latino middle school youth higher than other ethnic groups. One well-established precursor of adolescent ATOD use is psychosocial stress. The overall aim of this project is to test the efficacy of a culturally appropriate psychosocial program to prevent or reduce ATOD use among Latino immigrant youth. The intervention consists of: (1) encouraging parental involvement in child schooling, general parenting skills, and coping strategies ; (2) fostering child social emotional learning (SEL) through assigning a near-peer success coach to help develop critical thinking, problem solving, and goal setting skills; and (3) promoting positive peer affiliations through participation in regular activities that facilitate bonding to prosocial institutions.

The specific aims are:

(1) Evaluate the potential of the intervention to delay the initiation into or reduce ATOD use among Latino youth who are 1st to 2nd generation immigrants; and (2) Evaluate the intervention's ability to strengthen known protective factors against ATOD use among adolescents-specifically child personal agency and parent-child, peer, and school relationships.

The study's primary hypothesis is: The Unidos Se Puede program will delay initiation of ATOD use of current non-users and reduce use among current users.

To accomplish these aims, we propose an attention placebo randomized control trial. For this trial, we will recruit a sample of youth and their parents (N=120 dyads) from a random sample of Latino 6th and 7th grade students in Tulsa Public Schools. Those meeting the inclusion/exclusion criteria and agreeing to participate will provide baseline data before being randomly assigned to either the treatment or control condition (n=60 dyads each). Participants will be followed for 12 months post-baseline, during which time we will collect psychosocial measures annually near the end of each school year (May to June). The study will collect psychosocial measures from parents and youth.

ELIGIBILITY:
Inclusion Criteria:

* Self-identified as Latino (Hispanic),
* Spanish as the primary language spoken in home,
* Enrolled in 6th or 7th grade in public school at one of the target sites.

Exclusion Criteria:

* Currently undergoing mental health treatment,
* Not eligible to take end of year examinations due to cognitive limitations.

Ages: 12 Years to 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 240 (Estimated)
Dates: Start 2020-01-01 (Actual); Primary Completion 2023-08-31 (Estimated); Study Completion 2023-08-31 (Estimated)

PRIMARY OUTCOMES:
Change in past 30-day ATOD use (alcohol, tobacco, marijuana) | Baseline and 12 months post-baseline
  The ATOD outcome measure creates a single index of use by summing youth report of the frequency of their use during the past 30 days for each of the following substance: alcohol, tobacco and marijuana.

CONTACTS AND LOCATIONS:
Overall Officials: Ronald B Cox, PhD, Principal Investigator — Oklahoma State University
Locations (1):
- Oklahoma State University-Tulsa, Tulsa, Oklahoma, United States

IPD SHARING:
Plan to Share IPD: Undecided
The intent to share data with other researchers exists, however, a plan to do so has not yet been developed.

REFERENCES:
- [Derived] Cox RB, Washburn I, Greder K, Sahbaz S, Lin H. Preventing substance use among Latino youth: Initial results from a multistate family-based program focused on youth academic success. Am J Drug Alcohol Abuse. 2022 Jan 2;48(1):69-77. doi: 10.1080/00952990.2021.1981357. Epub 2021 Oct 28. PMID 34710334